CLINICAL TRIAL: NCT02596477
Title: A Phase 2 Randomized, Double-Blind, Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Vepoloxamer Injection, 22.5% (Sodium-Free) in Ambulatory Subjects With Chronic Heart Failure
Brief Title: Evaluation of Vepoloxamer in Chronic Heart Failure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated for administrative reasons not related to safety or efficacy
Sponsor: Mast Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MST-188-09
Record Dates: First submitted 2015-10-30; First posted 2015-11-04 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Heart Failure
Keywords: Heart failure
MeSH Terms: conditions — Heart Failure | interventions — Glucose; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vepoloxamer - Low dose (Experimental): Vepoloxamer injection administered intravenously 225 mg/kg over 3 hours
  Interventions: Drug: Vepoloxamer
- Vepoloxamer - High dose (Experimental): Vepoloxamer injection administered intravenously 450 mg/kg over 3 hours
  Interventions: Drug: Vepoloxamer
- 5% dextrose in water (D5W) (Placebo Comparator): D5W administered intravenously over 3 hours
  Interventions: Other: 5% dextrose in water

INTERVENTIONS:
Drug: Vepoloxamer
  Arms: Vepoloxamer - High dose; Vepoloxamer - Low dose
Other: 5% dextrose in water
  Other Names: D5W
  Arms: 5% dextrose in water (D5W)

SUMMARY:
The purpose of this study is to evaluate whether vepoloxamer can provide a blood chemical marker and functional benefit to damaged heart muscle cells. This will be evaluated by measurement of blood-based laboratory markers, exercise tolerance, and echocardiograms. In addition, the safety and blood levels of vepoloxamer in subjects with chronic heart failure will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 74
* Duration of documented heart failure >3 months
* On stable concomitant medication regimen ≥4 weeks
* Left ventricular ejection fraction ≤35%
* Systolic blood pressure ≥90 mmHg

Exclusion Criteria:

* Severe valvular stenosis or primary valvular regurgitation as the cause of heart failure
* History of myocardial infarction, coronary artery bypass graft surgery, or percutaneous intervention within the prior 3 months
* Estimated glomerular filtration rate ≤45 mL/min/1.73 m2
* Acutely decompensated heart failure within 1 month prior to the screening visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Number of subjects with a change in cardiac biomarkers ultra-high sensitive troponin I and NT-proBNP | Study Day 1 through Study Day 30
Number of subjects with a change in Six Minute Walk test | Study Day 1 to Study Day 30
Number of subjects with a change in Borg dyspnea index | Study Day 1 to Study Day 30
Number of subjects with a change in Minnesota Living with Heart Failure Questionnaire® | Study Day 1 to Study Day 30
Number of subjects with a change in left ventricular end diastolic volume index | Study Day 1 to Study Day 30
Number of subjects with treatment-related adverse events as assessed by CTCAE v 4.03 | Study Day 1 to Study Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Edwin L. Parsley, D.O., Study Director — Mast Therapeutics, Inc.
Locations (4):
- United States (2):
  - Research Center, Detroit, Michigan
  - Research Center, Tupelo, Mississippi
- Australia (2):
  - Research Center, Cardiff, New South Wales
  - Research Center, Melbourne, Victoria